CLINICAL TRIAL: NCT05648084
Title: To Investigate the Predictive Efficiency of Staging by Processing Tomography Images in Esophageal and Stomach Malignancies
Brief Title: Artificial Intelligence and Cancer Staging in Upper Gastrointestinal Malignancies
Status: Completed | Type: Observational
Sponsor: Sebahattin Celik MD (Other)
Responsible Party: Sponsor-Investigator, Sebahattin Celik MD, Associate Professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Other Study IDs: 2021-667-19/20210502
Record Dates: First submitted 2022-12-04; First posted 2022-12-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Esophageal and stomach cancers, which constitute cancers of the upper region of the digestive system, are cancers that are frequently observed and unfortunately have a low rate of cured patients. In these cases, the stage of cancer at diagnosis is very important for two reasons; First, the stage of the cancer is directly related to the survival time. Secondly, treatment is planned according to the stage. Different treatments are applied to patients at different stages. Currently, the TNM staging (Tumor, Lymph Node and Metastases) system is the accepted one worldwide. Despite many advanced technology tools used in staging (Computed Tomography, Magnetic Resonance Imaging, Endoscopic Ultrasonography), there are still difficulties in correct staging before surgery or before-after neoadjuvant therapy. Artificial intelligence techniques are increasingly used in the field of health, especially in the diagnosis and treatment of cancers. Obtaining cancer details in radiological images, which cannot be noticed by the human eye, by analyzing big data with the help of algorithms gave rise to the application area of "radiomics". It is stated that with Radiomics, there will be improvements in both the diagnosis and staging of cancers and, accordingly, in the treatment. While there are studies on the use of endoscopic methods with artificial intelligence for the early diagnosis of esophageal cancers, a limited number of studies have been conducted on stage estimation from radiological images. In particular, there are not enough studies on the investigation of changes in tumor size after chemotherapy with artificial intelligence and the estimation of staging. In this study, it was aimed to investigate the predictive efficiency of staging and the accuracy of the algorithm developed with artificial intelligence by processing tomography images in a region where esophageal cancers are endemic as a primary outcome and to evaluate the post-treatment mortality, morbidity rates and complication rates of the patients as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with esophageal cancer (adenocarcinoma or squamous cancer)
2. Being over 18 years old
3. Having a tomography image before or after chemotherapy.
4. Giving informed consent to participate in the study.
5. Having final pathological staging after surgery.

Exclusion Criteria:

1. Previous thoracic surgery.
2. Having a recurrent tumor
3. Inability to perform clinical staging due to technical reasons
4. Drawings cannot be made due to poor tomography quality.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: esophageal and stomach cancer patients over 18 years old diagnosed in 2 centers in van turkey, Van Training and Research Hospital and Van Yuzuncu Yıl University.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Artificial intelligence's sensitivity and accuracy to predict the stage of the cancer | 1 year
  to investigate the predictive efficiency of staging and the accuracy of the algorithm developed with artificial intelligence by processing tomography images in a region where esophageal cancers are endemic

SECONDARY OUTCOMES:
to evaluate the post-treatment mortality, morbidity rates and complication rates of the patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT05648084/Prot_SAP_000.pdf